CLINICAL TRIAL: NCT04870853
Title: Cardiovascular Events Among Adults Patients With Aggressive B-Cell Lymphoma Treated With Standard of Care Chimeric Antigen Receptor T Cell Therapy: A Single-Institution Experience
Brief Title: Cardiovascular Events Among Adults Patients With Relapsed or Refractory Aggressive B-Cell Lymphoma Treated With Standard of Care Chimeric Antigen Receptor T Cell Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-0120; NCI-2021-02675 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0120 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-04-12; First posted 2021-05-04 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Recurrent Aggressive B-Cell Non-Hodgkin Lymphoma; Recurrent Diffuse Large B-Cell Lymphoma; Recurrent High Grade B-Cell Lymphoma; Recurrent Primary Mediastinal (Thymic) Large B-Cell Lymphoma; Recurrent Transformed Follicular Lymphoma to Diffuse Large B-Cell Lymphoma; Refractory Aggressive B-Cell Non-Hodgkin Lymphoma; Refractory Diffuse Large B-Cell Lymphoma; Refractory High Grade B-Cell Lymphoma; Refractory Primary Mediastinal (Thymic) Large B-Cell Lymphoma; Refractory Transformed Follicular Lymphoma to Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (medical record review): Patients' medical records are reviewed retrospectively.
  Interventions: Other: Electronic Health Record Review

INTERVENTIONS:
Other: Electronic Health Record Review — Medical records reviewed

SUMMARY:
This study characterizes cardiac events following standard of care chimeric antigen receptor T cell therapy in patients with aggressive B-Cell Lymphoma that has come back (relapsed) or does not respond to treatment (refractory). The results from this study may allow a description of these events, their managements and outcome.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To characterize cardiac events following standard of Care (SOC) chimeric antigen receptor T (CAR-T) cell therapy in adult patients with relapsed/refractory aggressive B-cell lymphoma.

OUTLINE:

Patients' medical records are reviewed retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>= 18 years) with a diagnosis of aggressive B-cell lymphoma (such as transformed follicular lymphoma, diffuse large B-cell lymphoma, primary mediastinal B-cell lymphoma and high-grade B-cell lymphoma), who received standard of care (SOC) chimeric antigen receptor T (CAR-T) cell therapy at MD Anderson Cancer Center

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (>= 18 years) with a diagnosis of aggressive B-cell lymphoma, who received SOC CAR-T cell therapy at MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-04-02 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
To characterize cardiac events following standard of care (SOC) | through study completion, an average of 1 year
  Summary statistics will be provided for patient demographic, and clinical and biological variables. Continuous variables will be presented as mean +/- standard deviation or median (interquartile range), as appropriate based on normality, and categorical variables will be presented as percentages. Continuous data will be compared with the use of unpaired Student's t-tests or Wilcoxon rank-sum tests, as appropriate. Categorical data will be compared using the chi-square or the Fisher exact test. Univariate analyses will be performed to determine the association between the time of cytokine release syndrome symptoms and tocilizumab administration with cardiovascular events. Statistical significance will be defined using a 2-tailed p value =< 0.05.
To characterize cardiac events following chimeric antigen receptor T cell therapy (CAR-T) | through study completion, an average of 1 year
  Summary statistics will be provided for patient demographic, and clinical and biological variables. Continuous variables will be presented as mean +/- standard deviation or median (interquartile range), as appropriate based on normality, and categorical variables will be presented as percentages. Continuous data will be compared with the use of unpaired Student's t-tests or Wilcoxon rank-sum tests, as appropriate. Categorical data will be compared using the chi-square or the Fisher exact test. Univariate analyses will be performed to determine the association between the time of cytokine release syndrome symptoms and tocilizumab administration with cardiovascular events. Statistical significance will be defined using a 2-tailed p value =< 0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Raphael E Steiner, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States